CLINICAL TRIAL: NCT03985891
Title: A Randomized, Prospective Clinical Trial of Safety and Efficacy of JS001 Combined With Chemotherapy in Patients With Locally Advanced Colon Cancer (Perioperative Treatment)
Brief Title: The Efficacy of JS001 Combined With Chemotherapy in Patients With Locally Advanced Colon Cancer
Acronym: JSFOL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, zlkzengshan, Director，Chief Physician & Professor, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JSFOL--CC. V1.0
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Colonic Neoplasms; Chemotherapy Effect
Keywords: Colon cancer; PD-1; Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — toripalimab; Drug Therapy; Folfox protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS001 in combination with Folfox (Experimental): Patients who meet the enrollment criteria will receive Folfox(Oxaliplatin 85mg/m2 iv Day1; Leucovorin 400mg/m2 iv Day1; 5-FU 400mg/m2 iv bolus on Day1, then1200mg/m2/d x 2days(total 2400mg/m2 over 46-48 hours) iv continuous infusion repeat every 2 weeks) in combination with JS001 (3mg/kg, Q2W). Patients will receive 6 cycles treatment in pre-operation and same cycles after operation.
  Interventions: Drug: Anti-PD-1 Monoclonal Antibody JS001; Drug: Chemotherapy
- Folfox (Active Comparator): Patients who meet the enrollment criteria will receive Folfox(Oxaliplatin 85mg/m2 iv Day1; Leucovorin 400mg/m2 iv Day1; 5-FU 400mg/m2 iv bolus on Day1, then1200mg/m2/d x 2days(total 2400mg/m2 over 46-48 hours) iv continuous infusion repeat every 2 weeks). Patients need to receive 6 cycles treatment in pre-operation and same cycles after operation.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Anti-PD-1 Monoclonal Antibody JS001 — Anti-PD-1 monoclonal antibody combined with chemotherapy in patients with locally advanced colon cancer (perioperative treatment)
  Other Names: Toripalimab
  Arms: JS001 in combination with Folfox
Drug: Chemotherapy — Folfox
  Other Names: Folfox

SUMMARY:
Colon cancer is one of the most lethal malignancies, and colorectal cancer ranks the fifth leading cause of tumor-related mortality in China. FOLFOX is the recommended adjuvant/ neoadjuvant treatment for advanced colon cancer. JS001, as the first Chinese produced anti-PD-1 monoclonal antibody, has been approved by CFDA. This study aims to assess the safety and efficacy of JS001 in combination with FOLFOX as adjuvant/neoadjuvant treatment for patients with locally advanced colon cancer.

DETAILED DESCRIPTION:
Colon cancer is one of the most lethal malignancies, and colorectal cancer ranks the fifth leading cause of tumor-related mortality in China. FOLFOX is the recommended adjuvant/ neoadjuvant treatment for advanced colon cancer and it can improve the R0 resection rate, as well as reduce recurrence rate, but the overall responding rate is limited. Currently, immune checkpoint blocked (ICB) emerges as a promising approach in early colon cancer. JS001, as the first Chinese produced anti-PD-1 monoclonal antibody, has been approved by CFDA in melanoma. This study was designed as a prospective, randomized, controlled trial. Patients who meet the enrollment criteria will receive FOLFOX (Q2W) and JS001 (3mg/kg, Q2W) or only FOLFOX for neoadjuvant treatment 6 cycles in pre-operation and same treatment after operation, a total of six months. The assessment will be conducted in the 6th week and 13th week from the initiation date in the first cycle. The patients will be followed up for 5 years. The pCR rate, rCR rate, ORR, DFS, OS and Safety will be compared. This study aims to assess the safety and efficacy of JS001 in combination with FOLFOX as adjuvant/ neoadjuvant treatment for patients with locally advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced colon cancer patients diagnosed by pathologic biopsy，and the patients have defined indications for neoadjuvant chemotherapy by MDT group.
2. Patients may be available to undergo surgery.
3. Patient has at least 1 measurable lesions according to RECIST version 1.1;
4. Males and females aged ≥18 years.
5. ECOG score 0-1; Estimate life ≥1 year.
6. The main organs and bone marrow function are basically normal:

(1) Blood test White blood cell count (WBC)≥2000/mm^ 3; Absolute neutrophil count (ANC)≥1000/mm^ 3; Blood platelet count ≥100000/mm^ 3; Hemoglobin ≥9g/d; Serum creatine ≤ 2.0mg/dL; (2) Liver function Serum total bilirubin (TBIL) is within the normal range (normal range specified by the institution; Total bilirubin of Gilbert syndrome <3.0mg/dL); Serum Aspartate Transaminase (AST), serum Alanine Aminotransferase Transaminase (ALT) and alkaline phosphatase (ALP) ≤ 2.5 * upper limit of normal (ULN); International normalized ratio (INR) ≤1.5(or the patient is taking Warfarin for a long time, INR=2-3), and prothrombin time (PTT) ≤ULN (3) Pulmonary function Carbon Monoxide Diffusing Capacity (DLCO) ≥70% predictive OR; DLCO<70% and ≥55% , and the maximal oxygen consumption VO2 max ≥10L/min/Kg (cardiopulmonary assessment) or 6 minute walk experiment ≥500 meters; Patients with DLCO <55% are not included in this study; Pulse oximetry at rest or walking ≥92% (4) Cardiac function Baseline ECG showes no PR interval prolongation or atrioventricular block; 7. Patient and his/her mate must agree to follow instructions for method of contraception for the duration of the study period and within 6 months of the end of the study (eg. Intrauterine device, birth control pills or condoms); Serum or urine pregnancy test is negative within 7days prior to study enrollment and must be non-lactating; 8. Patients voluntarily joined the study, signed informed consent document, and were well compliant and able to be followed up with testers.

Exclusion Criteria:

1. Any previous active autoimmune disease (including any history of inflammatory bowel disease), or history of diseases to be treated with systemic steroids or immunosuppressive drugs(except for vitiligo patients）；
2. Use vaccines against infectious diseases (such as flu, chickenpox, etc.) within 4 weeks (28 days) of starting the study treatment;
3. Active systemic infection requiring treatment, positive detection of hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA);
4. A known positive history or positive test result of human immunodeficiency virus or acquired immunodeficiency syndrome (AIDS);
5. Patients with any severe and/or uncontrolled diseases, such as (1)unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmia；Patients with unsatisfactory blood pressure control (systolic blood pressure >140mmHg,diastolic blood pressure>90mmHg); (2) active or uncontrolled severe infection; (3) liver diseases such as cirrhosis, (4) decompensated liver disease, chronic active hepatitis; poor diabetes control (fasting blood glucose (FBG)> 10mmol/L); (5) urinary routine indicates urinary protein>or=++, and confirmed 24-hour urine protein quantitative >1.0g; (6) having a history of psychotropic substance abuse and being unable to quit or have mental disorders;
6. Pevious treatment with any anti-tumor treatment, including but not limited to chemotherapy, radiotherapy, immunotherapy (such as anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA-4 antibodies or any other antibodies that target the T cell co-regulatory pathway), etc; Tumor-related therapies or online anticancer drugs are currently being used; Anticoagulant is currently in use; Received major surgery in the past 3weeks;
7. Studies with previous malignancies, unless complete remission is achieved at least 2 years prior to the start of the study and no other treatment (subjects with basal cell carcinoma of skin and carcinoma in situ of cervix will not be excluded from the study);
8. History of previous interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, symptomatic interstitial lung disease, or evidence of any activepneumonia found on chest CT scans within 4 weeks prior to the first study drug treatment.
9. Immunosuppressive drugs were used within 2weeks prior to the first study drug treatment, excluding topical glucocorticoids, systemic glucocorticoids ≤ 10mg/day of prednisone or equivalent doses of other glucocorticoids;
10. Pregnant or lactating female;
11. Prisoners who are illegally imprisoned or compulsory for non-mental illness or physical (eg infectious disease) illness;
12. Patients with bleeding tendency (such as active gastrointestinal ulcers) or treatment with anticoagulants or vitamin K antagonists such as warfarin, heparin or the like;
13. A history of allergic reactions to the interventions;
14. According to the investigator's judgment, there are serious concomitant diseases that endanger the safety of the patient or affect the patient's completion of the study;

16. Has received a vaccine within 30 days prior to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-16 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | From the initiation date of first cycle to the date of operation, up to 5 months (each cycle is 2 weeks)
  Pathologic complete response rate
rCR rate | From the initiation date of first cycle to the date of operation, up to 5 months (each cycle is 2 weeks)
  Radiographic complete response rate
ORR | From the initiation date of first cycle to the date of operation, up to 5 months (each cycle is 2 weeks)
  Immunotherapy overall response rate

SECONDARY OUTCOMES:
DFS | From the initiation date of first cycle to the date of first documented progression, loss to follow up or death from any causes, whichever came first, up to 5 years (each cycle is 2 weeks)
  Disease-free survival
OS | From the initiation date of first cycle to the date of death from any causes or loss to follow up, whichever came first, up to 5 years (each cycle is 2 weeks)
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Shan Zeng, Ph.D, MD., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Shan Zeng, Changsha, Hunan, China